CLINICAL TRIAL: NCT04190355
Title: The Effect of Irrigant Types Used During Endodontic Treatment on Postoperative Pain: a Randomized Controlled Clinical Trial
Brief Title: The Effect of Irrigant Types Used During Endodontic Treatment on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Department of Endodontics, Principal Investigator, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11/29.05.2019
Record Dates: First submitted 2019-11-25; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain
Keywords: Root canal; irrigation; irrigant type; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group 1: 2 ml of 5.25% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Group 1: 2 ml of 5.25% Cloraxid gel/ distilled water will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation. The tip of the cannula will be adjusted to reach two-thirds of the working length.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5.25% NaOCl solution (Active Comparator): 5.25% NaOCl solution will be used as irrigation solution at every file change during root canal preperation
  Interventions: Other: Irrigant type; Drug: 5.25% NaOCl
- 5.25% Cloraxid gel/ distilled water (Active Comparator): 5.25% Cloraxid gel/ distilled water will be used as irrigation solution at every file change during root canal preperation
  Interventions: Drug: 5.25% Cloraxid gel/ distilled water

INTERVENTIONS:
Other: Irrigant type — The success of endodontic treatment is directly related to infection control. In successful endodontic treatment, it is necessary to perform an ideal irrigation both in order to gain a better understanding of the complex anatomical structure of the root canals and to increase the efficiency of the instruments and methods used during the canal preparation. Sodium hypochlorite (NaOCl) solution is the standard irrigation agent for cleaning and disinfection of root canal. In this study, the effect of NaOCI on postoperative pain using different uniforms will be evaluated.
  Arms: 5.25% NaOCl solution
Drug: 5.25% NaOCl — 5.25% NaOCl solution
  Arms: 5.25% NaOCl solution
Drug: 5.25% Cloraxid gel/ distilled water — 5.25% Cloraxid gel/ distilled water
  Arms: 5.25% Cloraxid gel/ distilled water

SUMMARY:
Chemomechanical preparation of the root canal system potentially results in extrusion of debris into the periradicular tissues. This debris is composed of hard tissue (dentin), soft tissue (inflamed or necrotic pulp tissues) and microbiota. Furthermore, the chemical adjuncts used during root canal disinfection may also extrude into the periradicular tissues. Extrusion of such materials results in postoperative pain, inflammation and and flare-up. There is evidence to demonstrate that most instrumentation techniques cause extrusion of debris, and that, severity of the inflammatory response depends on the amount of debris extrusion. Several factors may influence the debris extrusion during root canal preparation, including the instrument design, technique of use and irrigating agent used during preparation.Sodium hypochlorite (NaOCl) is the most commonly used root canal irrigant during root canal treatment. However, its cytotoxic effects when extruded into the periapical tissues is an issue of clinical concern. Thus, there has been a search for more biocompatible irrigants. One potential option, which has not been explored in detail, is the use of NaOCl, but in a gel form rather than a solution. NaOCl gel has similar effects on the dentin, as the solution form. Interestingly, greater dentinal tubule penetration depth has been reported for the gel form, compared to the solution. Previous studies have evaluated the effect of preparation techniques, the number of appointments and intracranial medicaments on postoperative pain during Endodontics treatment. There is no study evaluating the effect of different irritant type on PP. Therefore, this study will be evaluated the effect of different irritant type (gel or solution form of NaOCI) on postoperative pain.

DETAILED DESCRIPTION:
1. The study is planned to be performed on 104 patients who are aged between 18-45 years and who have no systemic disease and are diagnosed and followed up in Yüzüncü Yıl University Faculty of Dentistry, Department of Endodontics.
2. Patients who have been diagnosed with irreversible pulpitis will be included in the study group.
3. Patients with periapical lesions and incomplete apex development will not be included in the study group.
4. The access cavity will be prepared under local anesthesia.Working length of the canal will be determined as it ends in apical constriction, by using 15 k file with apex locater and periapical radiographs.
5. Preperation of root canals will be finished with ProTaperNext X3 instrument as standard and applied to each patient.
6. All patients will be randomly divided into two groups according to the irrigation protocol (G1: 5.25% NaOCI; G2: Chloraxid gel / distilled water) (n = 250).
7. Group 1: 2 ml of 5.25% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.

   Group 1: 2 ml of 5.25% Cloraxid gel/ distilled water will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation. The tip of the cannula will be adjusted to reach two-thirds of the working length.
8. Final irrigation procedure after canal preperation, 5 ml of 5.25% NaOCl solution, 5 ml of 17% EDTA solution, 5.25% NaOCl solution will be used respectively for both groups as standard.
9. After the final irrigation process, the root canals will be dried with sterile paper points, then they will be filled with sterile gutta-percha with lateral condensation technique by hand spredars. After root canal filling teeth will be restorated for coronal sealing.
10. After the treatment, the patients in both groups will be asked to report the pain levels at certain intervals (6th hour-24th hour-48th hour-72th hour-1st week) according to the VAS scale.
11. According to the questionnaires collected with patient feedbacks, the data will be analyzed and interpreted with statistical analysis ** (manwithney u-kruskall Wallis) in order to evaluate the pain levels after single visit root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Mandibular molar teeth that were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with calcified canals
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
VAS scala | up to 7 days
  PP will be assessed with a VAS after endodontic treatment. The VAS consisted of a 100-mm hor- izontal ruler with marks every 10 mm and no numbers except a 0 at the first part of the scale and a 10 in the last part of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Özlek, PhD, Study Chair — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Topcuoglu HS, Topcuoglu G, Arslan H. The Effect of Different Irrigation Agitation Techniques on Postoperative Pain in Mandibular Molar Teeth with Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2018 Oct;44(10):1451-1456. doi: 10.1016/j.joen.2018.06.008. Epub 2018 Aug 23. PMID 30144989